CLINICAL TRIAL: NCT03019887
Title: Correlation Between Cognitive Function and Relapse of Schizophrenia Regarding Dose Reduction in Patients Undergoing High-dose Antipsychotic Therapy
Brief Title: Correlation Between Cognitive Function and Relapse of Schizophrenia Regarding Dose Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juntendo University (Other)
Responsible Party: Principal Investigator, Ryota Ataniya, Clinician, graduate student, Juntendo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 673
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia Relapse
MeSH Terms: interventions — Haloperidol; Olanzapine; Quetiapine Fumarate; Aripiprazole; Paliperidone Palmitate; Methotrimeprazine; Perphenazine

ARMS (1):
- reduction group (Experimental): dose reduction of antipsychotics at a rate not exceeding 50mg chlorpromazine equivalent/week
  Interventions: Drug: reduction of risperidone, haloperidol, olanzapine, quetiapine, aripiprazole, paliperidone, levomepromazine, perphenazine

INTERVENTIONS:
Drug: reduction of risperidone, haloperidol, olanzapine, quetiapine, aripiprazole, paliperidone, levomepromazine, perphenazine

SUMMARY:
To reduce antipsychotics to under 1000mg in patients with schizophrenia taking more than 1000mg/day and to evaluate relationship between relapse and cognitive function.

DETAILED DESCRIPTION:
We attempted to reduce the dose of antipsychotics to ≤1000-mg chlorpromazine eq./day. The dose was gradually reduced at a rate of ≤50-mg chlorpromazine eq./week, and the reduction was discontinued if the subjects relapsed. The differences in baseline cognitive function were analyzed between the patients with no relapse and relapse groups.

ELIGIBILITY:
Inclusion Criteria:

* inpatients with a diagnosis of schizophrenia, and
* those in the chronic phase receiving mean daily antipsychotic doses exceeding 1000-mg chlorpromazine eq./day.

Exclusion Criteria:

* mental retardation,
* substance abuse or dependence,
* a history of major head trauma,
* serious medical or neurological disorders, or
* depot antipsychotic injections within the previous 3 months and electroconvulsive therapy within the previous 6 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takahashi Tadashi, Study Chair — Okada hospital; Mikiro Saito, Study Chair — Okada hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Reduction: patients who reduced dose of antipsychotics
Period: Overall Study
Arm/Group | Dose Reduction
Started | 139
Completed | 130
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Reduction Group: Group of patients with schizophrenia undergoing high-dose therapy (>1000-mg chlorpromazine eq./day) We attempted to reduce the dose of antipsychotics to ≤1000-mg chlorpromazine eq./day.
Arm/Group | Reduction Group
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 80
Region of Enrollment [Number; unit: participants]
  Japan | 130

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse
Description: The definition of relapse is as follows 1.50% or greater increase in total DIEPSS score, 2. an increase in the total PANSS score of 25% or more from baseline, 3. deliberate self-injury, 4. emergence of clinically significant suicidal ideation, 5. violent behavior resulting in clinically significant injury to another person or property damage.
Time Frame: One year after the baseline cognitive function test or three months after the end of dose reduction, whichever came first.
Population: patients with schizophrenia taking more than 1000 mg / day of antipsychotics, reduce their dose to less than 1000 mg
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Reduction
Number analyzed (Participants) | 130
Participants | 130

ADVERSE EVENTS:
Arm/Group | Dose Reduction
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 51/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Reduction (N=130)
increase in the total PANSS score from baseline (Psychiatric disorders) | 51
increase in total DIEPSS score (Psychiatric disorders) | 0
violent behavior (Psychiatric disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes